CLINICAL TRIAL: NCT01904071
Title: Ultrasound Guided Femoral (3 in 1) Nerve Block Versus Ultrasound Guided Fascia Iliacus Compartment Block Versus Standard Treatment for Pain Control in Patients With Hip Fractures in the Emergency Department
Brief Title: Ultrasound Guided Pain Control Versus Standard Treatment in Emergency Department HIP Fracture Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08/09/VA09
Record Dates: First submitted 2013-07-17; First posted 2013-07-22 (Estimated); Results first posted 2014-04-24 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2014-05

CONDITIONS: Hip Fracture
Keywords: Hip Fracture; Ultrasound; Nerve Block
MeSH Terms: conditions — Hip Fractures | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- UFNB (Experimental): Ultrasound guided 3 in 1 femoral nerve block: The UFNB was performed by first visualizing the femoral nerve in a transverse orientation just inferior to the inguinal ligament and lateral to the common femoral artery.
  Interventions: Procedure: UFNB (Ultrasound guided femoral nerve block)
- UFIB (Experimental): Ultrasound Guided Fascia Iliaca Compartment Block: For the UFIB, the two fascial planes, the fascia lata and the fascia iliaca, were sonographically visualized with the probe transverse to the thigh just inferior to the inguinal ligament and one-third of the distance from the anterior superior iliac spine to the pubic tubercle.
  Interventions: Procedure: UFIB (Ultrasound Guided Fascia Iliaca Compartment Block)
- IVMS (Active Comparator): IV Morphine: IV Morphine patients were also monitored for a minimum of one hour after they were given a second dose of IV morphine, 0.1 mg/kg, once the radiographs demonstrated fracture. The control group was also eligible to receive rescue analgesia of an additional 0.1 mg/kg of IV morphine, followed by repeat doses of 0.05 mg/kg
  Interventions: Drug: IVMS (IV Morphine)

INTERVENTIONS:
Procedure: UFNB (Ultrasound guided femoral nerve block) — Ultrasound Guided Femoral Nerve Block
  Arms: UFNB
Procedure: UFIB (Ultrasound Guided Fascia Iliaca Compartment Block)
  Arms: UFIB
Drug: IVMS (IV Morphine) — Intravenous Morphine
  Arms: IVMS

SUMMARY:
Hip Fracture (HFx) is a painful injury that is often treated in the Emergency Department (ED) with intravenous opiates. However, this class of medications may cause deleterious side effects. An alternative analgesic approach involves regional anesthesia. The investigators attempted to determine (1) whether ultrasound guided peripheral nerve blocks (UPNBs) could be safely performed in an ED setting, (2) whether UPNBs would be more effective than standard treatment in controlling pain from HFx and (3) which of two UPNBs was superior for pain relief.

A convenience sample of patients with an isolated HFx and a pain score > 5/10 were enrolled and randomized to one of three arms: (1) Ultrasound guided 3-in-1 femoral nerve block (UFNB), (2) Ultrasound guided fascia iliaca compartment block (UFIB), or (3) IVMS. Patients indicated their pain from 0 (no pain) to 10 (extreme pain).

DETAILED DESCRIPTION:
Hip fracture (HFx) is a painful orthopedic emergency that commonly presents to the Emergency Department (ED). There are approximately 320,000 HFx diagnosed annually in the United States, with this number expected to increase as the population ages. It has previously been shown that patients with pain from HFx are undermedicated while in the ED, particularly in overcrowded facilities. Current treatment for ED patients who are experiencing pain from acute HFx is often with intravenous morphine sulfate (IVMS). Morphine can have many undesirable side effects, but of particular concern are delirium, hypotension and respiratory depression. These complications may be accentuated in elderly patients and may necessitate increased patient monitoring and greater utilization of limited ED resources.An alternative to systemic opioid analgesia involves peripheral nerve blockade. Anesthesiologists frequently perform nerve blocks in the peri-operative and post-operative period to control pain in patients undergoing hip surgery. Traditionally, nerve stimulators were used to place the nerve block. However, ultrasonography is being used with increasing frequency to facilitate placement of these peripheral nerve blocks. As Emergency Physicians (EP) become more facile with the use of bedside sonography, ultrasound guided peripheral nerve blockade for HFx may be ideally suited for the ED environment, where one injection could control pain for many hours. The 3-in-1 femoral nerve block (FNB), in which anesthetic is injected adjacent to the femoral nerve but also affects the lateral femoral cutaneous and the obturator nerves, has been shown to be as effective as morphine for pain control of HFx in the ED. Sonographic guidance has been shown to increase the success rate of this block, decrease the time to analgesia, decrease the amount of local anesthetic needed to achieve adequate regional anesthesia, and decrease the incidence of inadvertent intravascular injection.

To date, there has been limited research describing the utilization of ultrasound guided femoral nerve blocks in an ED setting. Beaudoin et al. performed a feasibility study demonstrating that EP could effectively perform ultrasound guided femoral nerve blocks. Reid et al. found a significantly decreased time to complete analgesia when using sonographic guidance compared to an anatomic landmark technique. In this later study, anesthesia was assessed by checking skin sensation. Neither of these studies utilized a 3-in-1 nerve block, which may provide greater pain relief for patients with HFx.

The fascia iliaca compartment block (FIB) is also effective for treating pain due to HFx. It has been shown in the pediatric anesthesia and pediatric emergency medicine literature that it provides adequate analgesia, and may provide more effective analgesia than the FNB for femur fractures in children. Most of the studies describe the FIB being performed using a technique based on anatomic landmarks. One recent study described ultrasound guidance of the FIB (UFIB) increasing the efficacy of the sensory blockade (12). UFIB has not previously been studied in the ED setting.

We attempted to determine (1) whether ultrasound guided peripheral nerve blocks (UPNB) could be safely performed in an ED setting, (2) whether UPNB would be more effective than standard treatment in controlling pain from HFx in which a 2.5 unit decrease in pain scores was considered clinically significant, and (3) which of two UPNB was superior for pain relief.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking patients
2. ≥18 years of age
3. radiographic evidence of hip fracture
4. Patients must be awake, alert and oriented to time, place and person.
5. pain score of ≥ 5 in 10 point scale.

Exclusion Criteria:

1. cognitive deficits
2. allergic to amide-type local anesthetic or morphine
3. more injuries than just hip fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Dickman, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- [Background] Department of Health and Human Services, the Centers for Disease control, 2004
- [Background] Hwang U, Richardson LD, Sonuyi TO, Morrison RS. The effect of emergency department crowding on the management of pain in older adults with hip fracture. J Am Geriatr Soc. 2006 Feb;54(2):270-5. doi: 10.1111/j.1532-5415.2005.00587.x. PMID 16460378
- [Background] Fletcher AK, Rigby AS, Heyes FL. Three-in-one femoral nerve block as analgesia for fractured neck of femur in the emergency department: a randomized, controlled trial. Ann Emerg Med. 2003 Feb;41(2):227-33. doi: 10.1067/mem.2003.51. PMID 12548273
- [Background] Marhofer P, Schrogendorfer K, Wallner T, Koinig H, Mayer N, Kapral S. Ultrasonographic guidance reduces the amount of local anesthetic for 3-in-1 blocks. Reg Anesth Pain Med. 1998 Nov-Dec;23(6):584-8. doi: 10.1016/s1098-7339(98)90086-4. PMID 9840855
- [Background] Casati A, Baciarello M, Di Cianni S, Danelli G, De Marco G, Leone S, Rossi M, Fanelli G. Effects of ultrasound guidance on the minimum effective anaesthetic volume required to block the femoral nerve. Br J Anaesth. 2007 Jun;98(6):823-7. doi: 10.1093/bja/aem100. Epub 2007 May 3. PMID 17478453
- [Background] Marhofer P, Schrogendorfer K, Koinig H, Kapral S, Weinstabl C, Mayer N. Ultrasonographic guidance improves sensory block and onset time of three-in-one blocks. Anesth Analg. 1997 Oct;85(4):854-7. doi: 10.1097/00000539-199710000-00026. PMID 9322469
- [Background] Beaudoin FL, Nagdev A, Merchant RC, Becker BM. Ultrasound-guided femoral nerve blocks in elderly patients with hip fractures. Am J Emerg Med. 2010 Jan;28(1):76-81. doi: 10.1016/j.ajem.2008.09.015. PMID 20006206
- [Background] Reid N, Stella J, Ryan M, Ragg M. Use of ultrasound to facilitate accurate femoral nerve block in the emergency department. Emerg Med Australas. 2009 Apr;21(2):124-30. doi: 10.1111/j.1742-6723.2009.01163.x. PMID 19422409
- [Background] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Background] Wathen JE, Gao D, Merritt G, Georgopoulos G, Battan FK. A randomized controlled trial comparing a fascia iliaca compartment nerve block to a traditional systemic analgesic for femur fractures in a pediatric emergency department. Ann Emerg Med. 2007 Aug;50(2):162-71, 171.e1. doi: 10.1016/j.annemergmed.2006.09.006. Epub 2007 Jan 8. PMID 17210208
- [Background] Dalens B, Vanneuville G, Tanguy A. Comparison of the fascia iliaca compartment block with the 3-in-1 block in children. Anesth Analg. 1989 Dec;69(6):705-13. PMID 2589650
- [Background] Dolan J, Williams A, Murney E, Smith M, Kenny GN. Ultrasound guided fascia iliaca block: a comparison with the loss of resistance technique. Reg Anesth Pain Med. 2008 Nov-Dec;33(6):526-31. doi: 10.1016/j.rapm.2008.03.008. PMID 19258967
- [Result] Haines L, Dickman E, Ayvazyan S, Pearl M, Wu S, Rosenblum D, Likourezos A. Ultrasound-guided fascia iliaca compartment block for hip fractures in the emergency department. J Emerg Med. 2012 Oct;43(4):692-7. doi: 10.1016/j.jemermed.2012.01.050. Epub 2012 Apr 9. PMID 22494596
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043

RESULTS

PARTICIPANT FLOW:
Groups:
- UFNB: Ultrasound guided 3 in 1 femoral nerve block: The UFNB was performed by first visualizing the femoral nerve in a transverse orientation just inferior to the inguinal ligament and lateral to the common femoral artery.
  UFNB (Ultrasound guided femoral nerve block)
- UFIB: Ultrasound Guided Fascia Iliaca Compartment Block: For the UFIB, the two fascial planes, the fascia lata and the fascia iliaca, were sonographically visualized with the probe transverse to the thigh just inferior to the inguinal ligament and one-third of the distance from the anterior superior iliac spine to the pubic tubercle.
  UFIB (Ultrasound Guided Fascia Iliaca Compartment Block)
- IVMS: IV Morphine: IV Morphine patients were also monitored for a minimum of one hour after they were given a second dose of IV morphine, 0.1 mg/kg, once the radiographs demonstrated fracture. The control group was also eligible to receive rescue analgesia of an additional 0.1 mg/kg of IV morphine, followed by repeat doses of 0.05 mg/kg
  IVMS (IV Morphine)
Period: Overall Study
Arm/Group | UFNB | UFIB | IVMS
Started | 24 | 20 | 20
Completed | 24 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UFNB | UFIB | IVMS | Total
Number analyzed (Participants) | 24 | 20 | 20 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 82 (9.96) | 82 (7.74) | 85 (7.91) | 83 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 13 | 41
  Male | 7 | 9 | 7 | 23
Region of Enrollment [Number; unit: participants]
  United States | 24 | 20 | 20 | 64
Pain Score at Triage [Mean (Standard Deviation); unit: units on a scale] — Pain Scale: Scores range from 0 (no pain) to 10 (sever pain). A score of 5 is moderate pain.
  units on a scale | 5.17 (3.29) | 5.50 (3.99) | 6.98 (1.87) | 5.84 (3.23)

OUTCOME MEASURES:

1. Primary Outcome: Pain Score at 30 Minutes
Description: Pain Score at 30 minutes post-administration of pain control treatment. Pain Scale: Scores range from 0 (no pain) to 10 (sever pain). A score of 5 is moderate pain
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UFNB | UFIB | IVMS
Number analyzed (Participants) | 24 | 20 | 20
units on a scale | 1.94 (2.43) | 2.05 (2.61) | 5.13 (2.70)
Statistical Analysis 1: Comparison: UFNB vs UFIB vs IVMS; Test type: Superiority or Other; p < .0001, ANOVA

2. Secondary Outcome: Pain Score at 60 Minutes
Description: Pain score at 60 minutes post-administration of pain control treatment. Pain Scale: Scores range from 0 (no pain) to 10 (sever pain). A score of 5 is moderate pain
Time Frame: 60 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UFNB | UFIB | IVMS
Number analyzed (Participants) | 24 | 20 | 20
units on a scale | 2.58 (3.06) | 1.90 (2.38) | 4.40 (2.92)
Statistical Analysis 1: Comparison: UFNB vs UFIB vs IVMS; Test type: Superiority or Other; p < .05, ANOVA

3. Other Pre Specified Outcome: Pain Score at 120 Minutes
Description: Pain score at 120 minutes post-administration of pain control treatment. Pain Scale: Scores range from 0 (no pain) to 10 (sever pain). A score of 5 is moderate pain
Time Frame: 120 minutes
Population: Pain score was not obtained for one patient in the IVMS group at 120 minutes.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UFNB | UFIB | IVMS
Number analyzed (Participants) | 24 | 20 | 19
units on a scale | 2.65 (2.49) | 1.30 (1.89) | 4.00 (2.98)
Statistical Analysis 1: Comparison: UFNB vs UFIB vs IVMS; Test type: Superiority or Other; p < .005, ANOVA

4. Other Pre Specified Outcome: Pain Score at 240 Minutes
Description: Pain Score at 240 minutes post administration of pain control treatment. Pain Scale: Scores range from 0 (no pain) to 10 (sever pain). A score of 5 is moderate pain
Time Frame: 240 minutes
Population: Pain score was not obtained for one patient in the UFNB group at 240 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UFNB | UFIB | IVMS
Number analyzed (Participants) | 23 | 20 | 20
units on a scale | 3.15 (2.70) | 1.72 (1.98) | 4.83 (2.58)
Statistical Analysis 1: Comparison: UFNB vs UFIB vs IVMS; Test type: Superiority or Other; p < .001, ANOVA

5. Other Pre Specified Outcome: Pain Score at 480 Minutes
Description: Pain score at 480 minutes post administration of pain control treatment. Pain Scale: Scores range from 0 (no pain) to 10 (sever pain). A score of 5 is moderate pain
Time Frame: 480 minutes
Population: Pain scores were not obtained for 4 patients in the UFNB group, 3 patients in the UFIB group, and 3 patients in the IVMS group at 480 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | UFNB | UFIB | IVMS
Number analyzed (Participants) | 20 | 17 | 17
units on a scale | 3.20 (2.28) | 2.35 (3.07) | 3.74 (2.89)
Statistical Analysis 1: Comparison: UFNB vs UFIB vs IVMS; Test type: Superiority or Other; p = 0.342, ANOVA

ADVERSE EVENTS:
Time Frame: 240 minutes
Arm/Group | UFNB | UFIB | IVMS
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/24 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes